CLINICAL TRIAL: NCT03484533
Title: HIV Self-testing of Men to Increase Testing and Prevention Uptake Among Male Partners and Improve Postpartum ART Use in PMTCT B+ Programs in Uganda
Brief Title: HIV Self Testing of Male Partners of Women in PMTCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Harvard University (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Connie Celum, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00002257; R01MH113434 (NIH)
Record Dates: First submitted 2018-03-09; First posted 2018-04-02 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-06

CONDITIONS: ART Adherence; PMTCT; Linkage to Care; HIV; PrEP
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Women provided HIV Self-test kit (Active Comparator): Women will be given HIV self-test kits that they can then deliver to their male partners.
  Interventions: Behavioral: HIV self-test kit
- Women provided invitation letter-standard of care (Active Comparator): Women will be given an invitation letter for fast track HIV testing in the clinic that they will deliver to their male partners.
  Interventions: Behavioral: Standard of Care (invitation letters for fast-track HIV testing in the clinic)
- Male partners of women provided HIV self-test kit (Other): Male partners of women who were randomized to receive HIV self-test kits that could be delivered to their partner.
  Interventions: Behavioral: HIV self-test kit
- Male partners of women provided invitation letter (Other): Male partners of women who were randomized to receive an invitation letter - standard of care.
  Interventions: Behavioral: Standard of Care (invitation letters for fast-track HIV testing in the clinic)

INTERVENTIONS:
Behavioral: HIV self-test kit — Women who are randomized to the HIVST arm will be trained in the use and interpretation of HIVST, and given two oral fluid-based HIVST kits to use with or give to their partners, along with information about HIV testing and prevention and care services. We will offer men confirmatory testing regardless of their HIV test result through HIVST, counseling, and if negative, PrEP and if positive, ART.
  Arms: Male partners of women provided HIV self-test kit; Women provided HIV Self-test kit
Behavioral: Standard of Care (invitation letters for fast-track HIV testing in the clinic) — In the standard of care arm, we will give women invitation letters to deliver to their male partners to come to the ANC clinic for fast-tracked HIV testing. We will offer men counseling and if negative, PrEP and if positive, ART.
  Arms: Male partners of women provided invitation letter; Women provided invitation letter-standard of care

SUMMARY:
The investigators will conduct a randomized trial to evaluate whether provision of oral HIV self-test kits (HIVST) to HIV-positive pregnant women to provide to their male partner, increases the proportion of male partners who test and link to HIV care or prevention, compared to invitation letters for fast track testing. Pregnant women who are randomized to the arm with secondary distribution of HIVST to their male partners will be trained in the use and interpretation of HIVST, and given two oral fluid-based HIVST kits to use with or give to their partners, along with information about HIV testing and prevention and care services. The investigators will offer men confirmatory testing regardless of their HIVST result, counseling, and if negative, pre-exposure prophylaxis (PrEP) and if positive, antiretroviral therapy (ART). The investigators will provide counseling to minimize social harms of HIV self-testing, and additional counseling and referral to social support services when social harms occur. This project will address key challenges in PMTCT B+ programs, by evaluating innovative strategies to increase male partner's knowledge of their HIV status, disclosure, and involvement coupled with offering PrEP to HIV-negative men, ART to HIV-positive men, and encouraging post-partum ART continuation and adherence among HIV-positive women.

DETAILED DESCRIPTION:
Uganda has the fifth highest HIV burden globally and one of the highest fertility rates in Africa. Prevention of mother-to-child HIV transmission Option B+ (PMTCT B+) is national policy in Uganda. To maximize the prevention and clinical benefits of PMTCT B+, the challenges of low HIV testing by male partners and high rates of post-partum discontinuation of ART, insufficient adherence, and incomplete viral suppression need to be addressed. Women may be more likely to continue ART long-term and have higher adherence post-partum if their partner is tested, there is mutual disclosure of HIV status, and their partner takes ART or PrEP, depending on his status. Innovative approaches are needed to allow men to test in settings other than busy antenatal clinics, preferably where they have privacy, are comfortable and do not miss work. Innovative HIV testing technology -HIVST- could increase male partner's uptake of HIV testing, and prevention (PrEP) or ART (for all HIV-positive men). This study has been designed to address this gap through an enhanced PMTCT B+ program with HIV self-testing, and linkage to PrEP or ART, for male partners.

In a demonstration project the investigators recently completed among mutually disclosed East African HIV serodiscordant couples (the Partners Demonstration Project), integrated ART and PrEP delivery with time-limited PrEP for the HIV-negative partner as a 'bridge' until the HIV-positive partner was on ART for six months, and achieved viral suppression, was very acceptable, achieved very high uptake and adherence to ART and PrEP, and nearly eliminated HIV transmission. This protocol builds on that demonstration project by evaluating whether PMTCT outcomes are improved by increasing uptake of HIV testing and PrEP among HIV-negative men whose pregnant partner is HIV-positive. PrEP for HIV-negative male partners of HIV-positive pregnant women provides highly effective prevention benefits during an important 'season of risk' when men may have higher HIV acquisition risk from their partner if she is viremic (during the first few months after ART initiation, post-partum ART discontinuation or due to viral resistance), or from outside partners.

The investigators will conduct a randomized trial to evaluate whether provision of oral HIV self-test kits to HIV-positive pregnant women who are randomized to the HIVST arm, achieves higher uptake of their male partner's testing and linkages to HIV care and prevention among male partners, compared to invitation letters for fast track testing in the clinic (the standard of care). The investigators will recruit HIV-positive women ≥18 years accessing PMTCT B+ programs in Kampala, who have a male partner of unknown HIV status. Women will be randomized to the intervention (HIVST) or the control arm (invitation letters to deliver to partners to come for fast-track testing at the Antenatal Care (ANC) clinic where she receives care.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility

For all participants

* Able and willing to provide written informed consent
* Able and willing to provide adequate locator information for study retention purposes

For women

* Age ≥18
* Currently pregnant
* HIV-positive based on positive rapid HIV tests, according to national algorithm
* Not currently enrolled in an HIV treatment study
* Male partner not known to be HIV-positive or has not tested in the past 3 months

For men - In partnership with an HIV-positive pregnant woman in PMTCT B+

Exclusion criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — See eligibility criteria below
Enrollment: 736 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, MD MPH, Principal Investigator — University of Washington
Locations (1):
- Infectious Disease Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mujugira A, Nakyanzi A, Donnell D, Boyer J, Stein G, Bulterys M, Naddunga F, Kyomugisha J, Birungi JE, Ssendiwala P, Nsubuga R, Muwonge TR, Musinguzi J, Sharma M, Celum CL. Partner testing with HIV self-test distribution by Ugandan pregnant women living with HIV: a randomized trial. J Int AIDS Soc. 2023 Sep;26(9):e26156. doi: 10.1002/jia2.26156. PMID 37675834
- [Derived] Bulterys MA, Mujugira A, Nakyanzi A, Wyatt MA, Kamusiime B, Kasiita V, Kakoola GN, Nalumansi A, Twesigye C, Pisarski EE, Sharma M, Boyer J, Naddunga F, Ware NC, Celum CL. "Him Leaving Me - That is My Fear Now": A Mixed Methods Analysis of Relationship Dissolution Between Ugandan Pregnant and Postpartum Women Living with HIV and Their Male Partners. AIDS Behav. 2023 Jun;27(6):1776-1792. doi: 10.1007/s10461-022-03910-3. Epub 2022 Nov 8. PMID 36348192
- [Derived] Bulterys MA, Sharma M, Mugwanya K, Stein G, Mujugira A, Nakyanzi A, Twohey-Jacobs L, Ware NC, Heffron R, Celum C. Correlates of HIV Status Nondisclosure by Pregnant Women Living With HIV to Their Male Partners in Uganda: A Cross-Sectional Study. J Acquir Immune Defic Syndr. 2021 Apr 1;86(4):389-395. doi: 10.1097/QAI.0000000000002566. PMID 33148995

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data provided is for the women who were enrolled and randomized to the intervention of secondary distribution of HIV self-test kits to their male partner or standard of care delivery of invitation letter to their male partner to test for HIV at the clinic and for male partners who were consented later in the study.
Groups:
- HIV Self-test Kit: HIV self-test kit: We will conduct a randomized trial to evaluate whether provision of oral HIV self-test kits to HIV-positive pregnant women overcomes their male partners' reluctance to be tested in PMTCT clinics. Pregnant women who are randomized to the HIVST arm will be trained in the use and interpretation of HIVST, and given two oral fluid-based HIVST kits to use with or give to their partners, along with information about HIV testing and prevention and care services. We will offer men confirmatory testing regardless of their HIV test result through HIVST, counseling, and if negative, PrEP and if positive, ART.
- Invitation Letter-standard of Care: Standard of Care: In the standard of care arm, we will give women invitation letters to deliver to their male partners to come to the ANC clinic for fast-tracked HIV testing. We will offer men counseling and if negative, PrEP and if positive, ART.
- Male Partner (HIV Self-test Kit): Male partners of female participants randomized to receive the HIV self-test kit.
- Male Partner (Invitation Letter): Male partners of women randomized to receive the invitation letter
Period: Overall Study
Arm/Group | HIV Self-test Kit | Invitation Letter-standard of Care | Male Partner (HIV Self-test Kit) | Male Partner (Invitation Letter)
Started | 332 | 168 | 161 | 75
Completed | 291 | 146 | 54 | 25
Not Completed | 41 | 22 | 107 | 50

BASELINE CHARACTERISTICS:
Population: The baseline characteristics of the women who were enrolled and randomized to the intervention or control standard of care and their male partners who enrolled in the study.
Groups:
- HIV Self-test Kit: Female: HIV self-test kit: We will conduct a randomized trial to evaluate whether provision of oral HIV self-test kits to HIV-positive pregnant women overcomes their male partners' reluctance to be tested in PMTCT clinics. Pregnant women who are randomized to the HIVST arm will be trained in the use and interpretation of HIVST, and given two oral fluid-based HIVST kits to use with or give to their partners, along with information about HIV testing and prevention and care services. We will offer men confirmatory testing regardless of their HIV test result through HIVST, counseling, and if negative, PrEP and if positive, ART.
- Invitation Letter-standard of Care: Female: Standard of Care: In the standard of care arm, we will give women invitation letters to deliver to their male partners to come to the ANC clinic for fast-tracked HIV testing. We will offer men counseling and if negative, PrEP and if positive, ART.
- HIV Self-test Kit: Male Partner: HIV self-test kit: Male partners of randomized HIV-positive pregnant women who will be given oral fluid-based HIVST kits to use, along with information about HIV testing and prevention and care services. Men were offered confirmatory testing regardless of their HIV test result through HIVST, counseling, and if negative, PrEP and if positive, ART.
- Invitation Letter-standard of Care: Male Partner: Standard of Care: In the standard of care arm, male partners will be given invitation letters to come to the ANC clinic for fast-tracked HIV testing. We will offer men counseling and if negative, PrEP and if positive, ART.
- Total: Total of all reporting groups
Arm/Group | HIV Self-test Kit: Female | Invitation Letter-standard of Care: Female | HIV Self-test Kit: Male Partner | Invitation Letter-standard of Care: Male Partner | Total
Number analyzed (Participants) | 332 | 168 | 161 | 75 | 736
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [23 to 30] | 27 [23 to 31] | 32 [28 to 36] | 31 [27 to 36] | 27 [23 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 332 | 168 | 0 | 0 | 500
  Male | 0 | 0 | 161 | 75 | 236
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Uganda | 332 | 168 | 161 | 75 | 736

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Men Who Test for HIV in the Self-test Arm to Men Who Test for HIV in the Standard of Care Arm
Description: Evaluate whether the secondary distribution of HIV self-tests to enrolled male partners of HIV-infected Ugandan women in PMTCT B+ increases the proportion of male partners who test for HIV
Time Frame: Up to 12 months post-partum
Population: Overall 236 enrolled male partners tested for HIV
Measure: Number; unit: participants
Groups:
- HIV Self-test Kit: HIV self-test kit: The number of enrolled men who were given a oral fluid-based HIVST kits to use by their partner, along with information about HIV testing and prevention and care services.
  We will offer men confirmatory testing regardless of their HIV test result through HIVST, counseling, and if negative, PrEP and if positive, ART.
- Invitation Letter-standard of Care: Standard of Care: The number of enrolled men who received an invitation letters from their partner to come to the ANC clinic for fast-tracked HIV testing. We will offer men counseling and if negative, PrEP and if positive, ART.
Arm/Group | HIV Self-test Kit | Invitation Letter-standard of Care
Number analyzed (Participants) | 161 | 75
participants | 161 | 75

2. Primary Outcome: The Proportion of HIV-positive Men Who Initiate ART in the Self-test Arm to the Standard of Care Arm
Description: Evaluate whether the secondary distribution of HIV self-tests to male partners of HIV-infected Ugandan women in PMTCT B+ is associated with male partners uptake of ART if they test HIV-positive.
Time Frame: Up to 12 months post-partum
Population: There were 51 newly identified male partners living with HIV, between the two arms.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Self-test Kit | Invitation Letter-standard of Care
Number analyzed (Participants) | 38 | 13
Participants | 33 | 12

3. Primary Outcome: The Proportion of HIV-negative Men Who Initiate PrEP in the Self-test Arm to the Standard of Care Arm
Description: Evaluate whether the secondary distribution of HIV self-tests to male partners of HIV-infected Ugandan women in PMTCT B+ is associated with male partners uptake of PrEP if they test HIV-negative
Time Frame: Up to 12 months post-partum
Population: There were 185 male partners without HIV in the two arms.
Measure: Count of Participants; unit: Participants
Groups:
- HIV Self-test Kit: HIV self-test kit: The number of men who tested HIV negative via HIV self-test kit.
- Invitation Letter-standard of Care: The number of men who tested HIV negative via SOC.
Arm/Group | HIV Self-test Kit | Invitation Letter-standard of Care
Number analyzed (Participants) | 123 | 62
Participants | 72 | 41

4. Secondary Outcome: Viral Suppression at 12 Months Post-partum in HIV-infected Ugandan Women as Measured by Viral Load Testing
Description: Evaluate whether the secondary distribution of HIV self-tests to male partners of HIV-infected Ugandan women in PMTCT B+ is associated with effective post-partum viral suppression among HIV-infected Uganda women.
Time Frame: Up to 12 months post-partum
Population: There were 428 women with VL available at 12 months post-partum.
Measure: Count of Participants; unit: Participants
Groups:
- HIV Self-test Kit: The number of women randomized to the HIV self-test arm who had viral load data available at 12 months post-partum.
- Invitation Letter-standard of Care: The number of women randomized to the standard of care arm who had viral load data available at 12 months post-partum.
Arm/Group | HIV Self-test Kit | Invitation Letter-standard of Care
Number analyzed (Participants) | 284 | 144
Participants | 239 | 110

5. Secondary Outcome: The Acceptability of HIV Self-testing Among Pregnant Women Taking Part in PMTCT B+, and Their Male Partners
Description: HIV-infected pregnant women and their male partners, experiences, perspectives and views on HIV self-testing evaluated by an inductive content analytic approach conducted through qualitative interviews. This does not permit quantification of numbers of persons who endorsed particular themes. The main themes reported were 1. Women's fear about delivering HIV self-testing kits to their partner particularly if they had not previously disclosed their HIV status to their partner. 2. Variable strategies used by women to introduce HIV self-testing to their male partners. 3. Range of male partner responses to receiving an HIV self-testing kit. 4. Women's confidence in ability to interpret HIV self-test results for their partners. 5. Women's strategies to persuade their partners to link to HIV care or HIV PrEP.
Time Frame: Up to 12 months post-partum
Measure: Count of Participants; unit: Participants
Groups:
- Women in the HIV Self-test Secondary Distribution Arm: Women from the secondary distribution of HIV self-test kit arm were asked to participate in a in-depth interview about their experience.
- Male Partners: Male partners who were reached through the secondary distribution of HIV self-test were asked to participate in a in-depth interview about their experience.
Arm/Group | Women in the HIV Self-test Secondary Distribution Arm | Male Partners
Number analyzed (Participants) | 29 | 30
Participants | 29 | 30

ADVERSE EVENTS:
Time Frame: 12 months
Description: Social harms and pregnancy outcomes were recorded for the cohort, in addition to serious adverse events. We did not record death, SAEs, or Other AEs for male partners who were enrolled.
Arm/Group | HIV Self-test Kit: Female | Invitation Letter-standard of Care: Female
All-Cause Mortality (participants affected / at risk) | 2/332 | 2/168
Serious Adverse Events (participants affected / at risk) | 5/332 | 1/168
Other Adverse Events (participants affected / at risk) | 5/332 | 1/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV Self-test Kit: Female (N=332) | Invitation Letter-standard of Care: Female (N=168)
Hospitalization (Pregnancy, puerperium and perinatal conditions) | 5 (332) | 1 (168) — Hospitalization due to pregnancy complications.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV Self-test Kit: Female (N=332) | Invitation Letter-standard of Care: Female (N=168)
Social Harm (Social circumstances) | 5 (5) | 1 (1) — Social harm related to HIV disclosure by male partner testing

LIMITATIONS AND CAVEATS:
Pregnant women living with HIV (PWLHIV) were excluded if they reported intimate partner violence (IPV) in the prior year, results may not be generalizable. The HIV self-test (HIVST) arm allowed men to test at home, the proportion tested may be underestimated by the number who came to the clinic for confirmatory HIV testing and enrolment. Phone outreach may have biased the outcome of male partner testing to the null by increasing testing in the standard of care (SOC) arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT03484533/Prot_002.pdf
  • Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT03484533/SAP_003.pdf